CLINICAL TRIAL: NCT04011631
Title: The Efficacy and Safety of Internal Defibrillation: Evaluation of the iD-System™, One-Handed Disposable Internal Defibrillation System
Brief Title: Evaluation of the iD-SystemTM, One-Handed Disposable Internal Defibrillation System.
Acronym: iD-System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMART Clinical Products BV (Industry)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iD-System
Record Dates: First submitted 2019-06-17; First posted 2019-07-08 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Prospective interventional study with medical device.
Masking Description: The participants / patients treated in the study are blinded for the sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cardiac surgery (Experimental): All patients undergoing cardiac surgery at the Ziekenhuis Oost-Limburg, meeting all inclusion and no exclusion criteria, are asked to participate in the investigation.
  Interventions: Procedure: Internal defibrillation during cardiac surgery, using the iD-system

INTERVENTIONS:
Procedure: Internal defibrillation during cardiac surgery, using the iD-system — When ventricular fibrillation of ventricular tachycardia occurs during surgery, the iD-Paddle will be applied directly to the heart. A maximum of 4 shocks are delivered to the heart to restore normal sinus rhythm. If 4 shocks are not successful standard operating procedure will be enable conform hospital protocol.

SUMMARY:
The main aim is to evaluate the safety and efficacy of the iD-System™, One-handed Disposable Internal Defibrillation System The device is made for manual defibrillation during intra-thoracic procedure, by transferring a shock from a defibrillation device to the patient's heart, in combination with the iD-Electrode. The device will be used when the patient reaches a stage of ventricular fibrillation or rapid ventricular tachycardia during cardiac surgery.

DETAILED DESCRIPTION:
The main aim is to evaluate the safety and efficacy of the iD-System™, One-handed Disposable Internal Defibrillation System The device is made for manual defibrillation during intra-thoracic procedure, by transferring a shock from a defibrillation device to the patient's heart, in combination with the iD-Electrode. The device will be used when the patient reaches a stage of ventricular fibrillation or rapid ventricular tachycardia during cardiac surgery.

In case ventricular fibrillation occurs and the iD-system is not effective to restore the sinus trythm, the conventional approach with use of the two paddels spoons will be performed immediately.

the following will be assessed:

* Ease of use of the device
* Safety of the device
* Efficacy of the device

ELIGIBILITY:
Inclusion Criteria:

* All races and ethnicity (>18 years)
* Written informed consent form (ICF) has to be obtained from the patient.
* Elective surgery: cardiac surgery on pump (CPB)

  * Coronary artery bypass surgery
  * Heart valve repair and/or replacement

    * Mini sternotomy
    * Median sternotomy
  * Redo surgery

Exclusion Criteria:

* Patients without cardiopulmonary bypass (referred to as heart-lung machine or pump)
* Emergency surgery without a sufficient amount of time to explain and ask for ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Beran, Dr., Principal Investigator — Anesthesiologist
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A cohort of 100 successive patients undergoing major cardiac surgery from 3 September 2018 to 6 February 2019 are included.
Period: Overall Study
Arm/Group | Patients With Cardiac Surgery
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Cardiac Surgery
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Skin Symptoms
Description: Safety of the iD-system will be evaluated to assess if there are skin symptoms to the electrode by confirming if irritation is visible on the back of the patient after removal of the iD elektrode or not. For the more subjects the irritation will be visible, the worse will be the safety of the iD-elektrode.
Time Frame: During intra-thoracic procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cardiac Surgery
Number analyzed (Participants) | 100
Participants | 0

2. Primary Outcome: Number of Patients With Increased Troponin-t Level Classified as Adverse Event
Description: Safety of the iD-system will be evaluated via troponine measurement to assess myocardial injury. Troponine will be measured at 4, 8, 16, 24 and 36 hours post-surgery and will be reported in ng/L. A significant increase of the troponine value during these different time points indicates myocardial injury. The investigator will evaluate every case to assess if it is an Adverse Event or not.
Time Frame: During intra-thoracic procedure till 36 hours post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cardiac Surgery
Number analyzed (Participants) | 100
Participants | 5

3. Primary Outcome: Number of Patients Where the iD-System TM Fails
Description: Efficacy of the the iD-System will be evaluated to assess a successful restoration of the sinus rythm by counting the number of failed attempts to defibrillate which were attributable to device malfunction. This will be captured by a questionnaire, to be completed by the investigator after the surgery. A maximum of 4 shocks can be applied. If the normal arterial hearth rhythm cannot be restored after 4 shocks with the iD-System, conversion to the conventional system occurs.
Time Frame: During intra-thoracic procedure
Population: Of the 100 patients that required cardiac surgery, 11 required defibrillation.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cardiac Surgery
Number analyzed (Participants) | 11
Participants | 1

4. Primary Outcome: Ease of Use of the iD-System as Assessed Via Investigator Questionnaire
Description: Ease of use of the iD-System will be evaluated by a questionnaire, to be completed after the procedure. The following items will be assessed:
  * adherence of the iD-Electrode to the patient's back
  * positioning of the iD-Padde for maximal contact with the heart
  * working length of the following cables: iD-Electrode,iD-Paddle and the iD-SMART Cable
  The questionnaire will consist of 16 questions, each addressing a specific topic of the ease of use, to be scored by the investigator from 1 to 5.
  1= very poor, 2= poor, 3= neutral, 4= sufficient, 5= excellent
  The higher the total score, the better the outcome of the 'ease of use' evaluation.
Time Frame: During intra-thoracic procedure
Population: The initial connection of the iD-system was done in all (100) cases. Paddles were tested in 98 percent.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cardiac Surgery
Number analyzed (Participants) | 100
Participants
  number of patients where connection was not successful | 0
  number of patients with visible skin irritation | 0
  number of patients wher cable length was considered not long enough: number analyzed (Participants) | 98
  number of patients wher cable length was considered not long enough | 91
  number of patients with connection problems with the defibrillator: number analyzed (Participants) | 98
  number of patients with connection problems with the defibrillator | 0
  number of patients where the contact surface was not sufficient: number analyzed (Participants) | 98
  number of patients where the contact surface was not sufficient | 0
  number of patients where th paddle was too large: number analyzed (Participants) | 98
  number of patients where th paddle was too large | 0
  number of patients with any other problems: number analyzed (Participants) | 98
  number of patients with any other problems | 0

ADVERSE EVENTS:
Time Frame: SAEs were reported in patients until discharge from ICU, up to 48 hours.
Arm/Group | Patients With Cardiac Surgery
All-Cause Mortality (participants affected / at risk) | 3/100
Serious Adverse Events (participants affected / at risk) | 6/100
Other Adverse Events (participants affected / at risk) | 16/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Cardiac Surgery (N=100)
Stroke (Vascular disorders) | 1 (1) — day 2 after complex cardiac surgery: stroke due to occlusion left middle cerebral artery. Extensive infacrction with cerebral herniation. No surgical treatment. outcome: death
Acute Kidney Injury (AKI) (Renal and urinary disorders) | 1 (1) — Prolonged ICU length of stay with AKI, low cardiac output syndrome and ventilator-associated pneumonia. outcome: recovered
Bleeding (Vascular disorders) | 1 (1) — D0: CABG + Mitral Valve plasty (patient known with cardiomyopathy + reduced LV function)) D1: revision for acute massive bleeding D6: revision for bleeding: vasoplegia + cardiogenic shock, resistent to therapy outcome: death Study device not used
Multi Organ Failure (MOF) (General disorders) | 1 (1) — (D0 redo CABG + mitral valve replacement) Patient known with reduced LVEF and MI D1: Difficult weaning CPB due to LV failure and vasoplegia R/IABP In ICU deterioration of cardiogenic shock and MOF. outdome: death Study device not used
Atrial Fibbrillation (Cardiac disorders) | 1 (1) — Atrial fibrillation, not well tolerated, loss of cardiac output resuscitation (CPR) , reintubation and ventilation reurn of spontaneous circulation within 10 minutes outcome: resolved
Status Epilepticus (Nervous system disorders) | 1 (1) — Difficult weaning post-op CABG/AVR. EEG revealed status epilepticus (patient known with epilepsy) outcome: ongoing
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Cardiac Surgery (N=100)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Multiple Organ Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Ventilator-associated pneumonia
Elevated Troponin-T level (Cardiac disorders) | 5 (5)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) — followed by ICU acquired weakness
Acute Kidney Injury - Failure (Renal and urinary disorders) | 1 (1) — known chronic renal failure
Diplopia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — pituitary adenoma
Trombopenia (Blood and lymphatic system disorders) | 1 (1)
Subdural hematoma (Vascular disorders) | 1 (1)
Delirum (General disorders) | 1 (1)
Decreased kidney function (Renal and urinary disorders) | 1 (1)
Endocarditis (Cardiac disorders) | 1 (1)
Ischemic stroke (Vascular disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT04011631/Prot_SAP_000.pdf